CLINICAL TRIAL: NCT03701412
Title: Prevalence of Cerebral Micro-bleeds in Patients With Cerebrovascular Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salah A Sabreen, principle investigator, Assiut University
Other Study IDs: POCMIPWCVS
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Cerebrovascular Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MRI — MRI brain

SUMMARY:
Cerebral microbleed (CMB) refers to small, round dark-signal lesions detected by T2*-weighted or gradient-echo (GRE) magnetic resonance imaging (MRI) ..CMBs were introduced to stroke physicians in the late 1990s and early 2000s after development of MRI techniques sensitive to paramagnetic effects The clinical significance of CMBs has been actively investigated, especially in the stroke field and more recently in studies on cognitive impairment, vascular dementia and later developement of cerebral hge ..Histological investigation has shown that CMBs are tiny foci containing hemosiderin-laden macrophages and abnormal microvessels . Clinical cases with frank symptoms caused by CMBs are uncommon, Because CMBs are manifestations of focal extravascular leakage of blood components, however, investigators have suggested that accumulation of CMBs reflects a bleeding-prone status in individuals with an elevated risk of cerebral hemorrhage. Clinical studies have found strong associations between CMBs and chronic hypertension and low cholesterol levels and between the proximity and volume of CMBs and those of subsequent intracerebral hemorrhage (ICH) . studies have found that CMBs are linked to subsequent hemorrhagic stroke in stroke survivors,and suggested that CMBs are related to antithrombotic-related hemorrhage.

DETAILED DESCRIPTION:
Cerebral microbleed (CMB) refers to small, round dark-signal lesions detected by T2*-weighted or gradient-echo (GRE) magnetic resonance imaging (MRI). CMBs were introduced to stroke physicians in the late 1990s and early 2000s after development of MRI techniques sensitive to paramagnetic effects The clinical significance of CMBs has been actively investigated, especially in the stroke field and more recently in studies on cognitive impairment, vascular dementia and later developement of cerebral hge ..Histological investigation has shown that CMBs are tiny foci containing hemosiderin-laden macrophages and abnormal microvessels .

Clinical cases with frank symptoms caused by CMBs are uncommon, Because CMBs are manifestations of focal extravascular leakage of blood components, however, investigators have suggested that accumulation of CMBs reflects a bleeding-prone status in individuals with an elevated risk of cerebral hemorrhage. Clinical studies have found strong associations between CMBs and chronic hypertension and low cholesterol levels and between the proximity and volume of CMBs and those of subsequent intracerebral hemorrhage (ICH) . studies have found that CMBs are linked to subsequent hemorrhagic stroke in stroke survivors,and suggested that CMBs are related to antithrombotic-related hemorrhage.

Clinical implications of cerebral microbleeds The increased of cerebral hemorrhage associated with the presence of CMBs may allow prediction of hemorrhagic transformation after ischemic stroke. An earlier report suggested that hemorrhagic transformation after thrombolysis was associated with the presence of CMBs.

Considerable interest also exists in utilizing detection of CMBs to estimate the risks of hemorrhagic complications in patients on antithrombotic treatment. , CMBs were found to be more frequent and extensive in patients with double antiplatelets-associated ICH.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as ischemic CVS or Transient ischemic attack admitted to Assuit University Hospital or visiting outpatient clinic.
* Old stroke patients on double antiplatelet therapy for duration more than 3 months
* old stroke patients on anticoagulants.

Exclusion Criteria:

* Patients with blood diseases hepatic and renal patient. Patients with cerebral hemorrhage.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients fulfilling previous criteria will undergo T2*-weighted or gradient-echo (GRE) magnetic resonance imaging (MRI) for detection of microbleeds,
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
analyse Risk factors responsible for development of cerebral micro bleeds. | 1 year
  All patients will undergo T2*-weighted or gradient-echo (GRE) magnetic resonance imaging (MRI) for detection of micro bleeds

IPD SHARING:
Plan to Share IPD: Undecided